CLINICAL TRIAL: NCT06856759
Title: Study on the Safety, Tolerability, and Preliminary Efficacy of Single Intrathecal Injection of AAV-MECP2 in the Treatment of Rett Syndrome
Brief Title: Single-Dose AAV-MECP2 Safety/Tolerability and Efficacy in Rett Syndrome
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-433A01
Record Dates: First submitted 2024-12-29; First posted 2025-03-04 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; AAV-MECP2; Single intrathecal injection; Safety; Tolerability; Preliminary efficacy
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose study on single Intrathecal injection of AAV-MECP2 for the treatment of Rett syndrome (Experimental): We plan to explore two target doses, with 5 subjects enrolled in dose 1 and 3 subjects enrolled in dose 2, to evaluate the safety, tolerability, and preliminary efficacy of a single intrathecal injection of AAV-MECP2 in the treatment of RTT.
  Interventions: Genetic: Intrathecal injection of AAV-MECP2 for the treatment of Rett syndrome

INTERVENTIONS:
Genetic: Intrathecal injection of AAV-MECP2 for the treatment of Rett syndrome — For Dose 1, the first 5 subjects will be enrolled in the trial in sequence, with one patient completing the administration and no significant dose limiting toxicity (DLT) observed during a one month follow-up. The latter subject will be enrolled in the trial medication.
  Once the fifth subject in Dose 1 completes the administration and no significant DLT is observed after a follow-up period of at least two weeks, the study dose can be escalated to a higher level.
  For Dose 2, the 3 subjects will be enrolled in the trial in sequence, with one patient completing the administration and no significant DLT observed during a one month follow-up. The latter subject will be enrolled in the trial medication.
  DLT definition: see Study Description.

SUMMARY:
Rett syndrome (RTT) is a serious neurodevelopmental disorder that has a significant impact on patients and their families. Patients suffer from severe social dysfunction and poor quality of life, and there is currently no effective treatment available. The MECP2 functional loss mutation is the clear pathogenic factor. In recent years, gene therapy has been applied in neuromuscular diseases such as SMA and has achieved good safety and effectiveness. Professor Qiu Zilong's self-developed AAV-MECP2 gene therapy product for RTT was found to significantly improve disease symptoms in RTT model mice, and demonstrated good safety in heath injection testing in monkeys. The dose exploration study of AAV-MECP2 initiated by our researchers is a multicenter, single arm, single intrathecal injection. The plan is to explore two target doses, with 5 subjects enrolled in dose 1 and 3 subjects enrolled in dose 2, to evaluate the safety, tolerability, and preliminary efficacy of single intrathecal injection of AAV-MECP2 in the treatment of RTT.

DETAILED DESCRIPTION:
Research background:

Rett syndrome (RTT) is a congenital neurodevelopmental disorder that mainly affects women. Its typical clinical manifestations include cessation or even regression of neural development from 6-18 months after birth, loss of acquired skills such as cognition, language ability, and hand function, often accompanied by stereotyped hand movements, abnormal respiratory rhythms, seizures, and anxiety disorders. RTT is a rare disease with a incidence rate of about 1/10000-15000, which is estimated to account for more than 10% of female intellectual disability. It has a great impact on patients and their families, with severe damage to their social functioning and a very poor quality of life.

Approximately 90-95% of typical RTT patients and 40-50% of atypical RTT patients have detected abnormalities in the methylation CpG binding protein 2 (MeCP2) encoding gene, as well as mutations or deletions in the MECP2 gene. The human MECP2 gene is located at Xq28, and its encoded protein methylated CpG binding protein 2 is a member of the methylation domain family. It is a transcription inhibitory factor that regulates RNA splicing and is a key epigenetic regulator in the brain, affecting neural function. In animal experiments, it was found that Mecp2 deficient mice showed significant improvement in RTT symptoms after receiving Mecp2 protein supplementation through genetic engineering technology.

In recent years, the success of gene therapy in neuromuscular diseases such as spinal muscular atrophy (SMA) has demonstrated the feasibility of applying gene therapy technology in the human body. Since 2023, TAYSHA (intrathecal administration) and Neurogene (intracerebroventricular administration) have respectively initiated gene therapy clinical trials for Rett syndrome. Currently, 2 adult RTT patients and several pediatric RTT patients have completed dosing. At doses ≤1.0×10^15 vg/person, the treatment continues to demonstrate a favorable safety profile with no serious treatment-related adverse events reported. No signs or symptoms indicative of MECP2 overexpression induced toxicity have been observed. Neurogene reported a serious adverse event (SAE) in the 3rd subject receiving a higher dose (3×10^15 vg/person) via intracerebroventricular administration, resulting in patient death. This suggests that excessive dosing may lead to severe adverse reactions.

Professor Qiu Zilong, a senior researcher at the Songjiang Research Institute of Shanghai Jiao Tong University School of Medicine, has been conducting long-term research on RTT. In 2012, it was discovered that MECP2 regulates neuronal synaptic homeostasis plasticity; In 2014, it was discovered that MECP2 regulates microRNA splicing processing; Established MECP2 transgenic crab eating monkey animal model in 2016; In 2019, the neural mechanism of MECP2 mice was identified and gene editing intervention therapy was attempted; Establish a MECP2 mutant mouse AAV gene therapy technology roadmap in 2022 and apply for an invention patent. The independently developed AAV-MECP2 significantly prolonged the lifespan of MECP2 knockout mice in lateral ventricle injection experiments, and the therapeutic effect of AAV-MECP2 with CAG promoter was significantly better than similar products. The safety and efficacy of intrathecal administration in monkey have been tested for 3 months, and blood routine, blood biochemistry, and immune factor indicators have all shown good safety.

In summary, RTT is a serious neurodevelopmental disorder that poses great harm to patients, and there is currently no effective treatment method. The clinical trial initiated by our researchers aims to evaluate the safety, tolerability, and preliminary effectiveness of AAV-MECP2 in the treatment of Rett syndrome through a single intrathecal injection, which has important medical and social value. The safety and efficacy of intrathecal administration have been tested for 3 months, and blood routine, blood biochemistry, and immune factor indicators have all shown good safety.

Research overview:

Overall research design:

A multicenter, single arm, single intrathecal dose exploration study of AAV-MECP2 initiated by researchers aims to explore two target doses, with 5 subjects enrolled in dose 1 and 3 subjects enrolled in dose 2, to evaluate the safety, tolerability, and preliminary efficacy of single intrathecal injection of AAV-MECP2 in the treatment of RTT.

Study population:

Children aged 4-10 years who have been diagnosed with RTT through consultation in Guangzhou Women and Children's Medical Center.

Test location:

Guangzhou Women and Children's Medical Center.

Exit criteria midway:

Family members can still withdraw from the study after obtaining informed consent.

Criteria for detachment/exclusion:

i. The patient needs to adjust the treatment medication used during the study period;

Ii. During the study, the use of drugs/treatments that are prohibited from the study is required: During the study, the following concomitant drugs/treatments are prohibited:

Drugs used to treat muscle disorders or neurodegenerative diseases (excluding antiepileptic drugs).

A drug used to treat diabetes. Immunosuppressants (such as glucocorticoids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab, etc.) were started within 3 months before enrollment.

After being enrolled in the study, a rehabilitation treatment plan that had never been carried out before is initiated.

iii. Unable to attend treatment at the hospital in one week according to the established medication plan; iv. After communication and coordination of time, the project evaluation cannot be completed; v. If any adverse events, laboratory abnormalities, or other medical conditions occur during the study period, and appropriate measures are taken, the researchers believe that continuing the trial may increase the risk for the subjects.

Number of participants and grouping method:

There will be 8 participants in the injection group. For Dose 1, the first 5 subjects will be enrolled in the trial in sequence, with one patient completing the administration and no significant dose limiting toxicity (DLT) observed during a one month follow-up. The latter subject will be enrolled in the trial medication.

Once the fifth subject in Dose 1 completes the administration and no significant DLT is observed after a follow-up period of at least two weeks, the study dose can be escalated to a higher level. For Dose 2, the 3 subjects will be enrolled in the trial in sequence, with one patient completing the administration and no significant DLT observed during a one month follow-up. The latter subject will be enrolled in the trial medication.

DLT definition: Any of the following events (graded according to NCI CTCAE V5.0) that occur within 30 days after administration and are determined by the researcher to be possibly or definitely related to AAV-MECP2 (see 4.2 Adverse Event Severity): ≥ Grade 3 adverse event; Level 3 laboratory abnormalities persist for ≥ 7 days with necessary medical intervention; Level 4 laboratory abnormality.

Experimental drug:

Experimental medication: AAV-MECP2; Active ingredient: recombinant AAV gene therapy vector containing neuron specific promoter (CAG) driven MECP2; Accessories: 4-hydroxyethylpiperazine ethanesulfonic acid, potassium chloride, sodium chloride, calcium chloride, glucose, poloxamer F68, and injection water; Dosage form: Intrathecal injection; Appearance: Colorless and transparent liquid; Specification: Independently packaged penicillin bottle, with a titer of 2 × 10^14 vg/mL and a volume of 0.5 mL; Administration route: intrathecal injection; Administration frequency: 1 time.

Research Steps and Methods:

1. Intervention method: AAV-MECP2, two exploratory doses (dose 1, dose 2, detailed below), single intrathecal injection;

   Drug dosage:

   The dose exploration rules have evolved from the traditional "3+3 design". The two pre-set dose levels for this study are: dose 1 (7 × 10^14 vg/person); dose 2 (1.0 × 10^15 vg/person).

   The two pre-set dose levels in this study are the initial dose level of dose 1 and a higher dose level of dose 2. During the research process, it is possible to explore a dose level below dose 1 or an intermediate dose between dose 1 and dose 2 based on accumulated safety and efficacy data, subject to SRC approval.

   At dose 1 level, 5 subjects were enrolled first, and then during the DLT observation period, the number of subjects who developed DLT among the 5 subjects was observed. Based on the number of subjects observed to have DLT, decide whether to increase to the next dose group, maintain the current dose group, or decrease to a lower dose group.
   1. If none of the 5 subjects enrolled in dose 1 develop DLT or only one subject develops DLT, the dose can be increased to a higher dose group. If 1 of the 3 subjects enrolled in dose 2 develop DLT, the trial should be stopped.
   2. If 2 out of the 5 subjects enrolled in dose 1 develop DLT, the administration to new subjects will be suspended until SRC makes a decision; At this point, after a comprehensive evaluation of the current safety and efficacy data, SRC will provide one of the following three resolutions: ① reduce the dose to a lower dose and enroll three assessable subjects; ② Add 3 additional assessable subjects to the current dose; ③ Stop the experiment.

   SRC stands for Safety Review Committee, responsible for reviewing safety data of subjects, composed of researchers and collaborating medical monitors. During the research process, SRC is responsible for protecting the safety of the subjects, and its responsibilities are as follows:

   Review the safety issues of each participant; Regularly review safety data while the subjects continue to receive study treatment; Evaluate whether it is necessary to expand the number of subjects in each stage and whether it is possible to proceed to the next dose stage, including dose escalation or dose reduction; Keep research data and results confidential.
2. Drug management:

For all received research intervention products, the researcher or designated personnel must confirm that appropriate temperature conditions are maintained during transportation, and any inconsistencies have been reported and resolved before using the research intervention products. This research product is packaged in penicillin bottles and transported by dry ice. After receiving it, the research center stores it at -75 ± 15 ℃.

Only enrolled subjects can receive research interventions, and only authorized research center staff can provide or administer research interventions. All research interventions must be stored in a safe, environmentally controlled, and monitored (manually or automatically) area according to the indicated storage conditions, and only researchers and authorized research center staff have access to the area.

The researcher or drug manager of the research center shall count and verify the research intervention products and maintain relevant records (i.e. receiving and verifying records and final disposal records).

Research evaluation:

The research program and its schedule can be found in the 'Research Schedule'. This table lists all evaluations and uses "X" to represent the evaluations performed at each visit. If the subject is unable to go to the trial center due to special reasons, the subject or their legal representative may contact the staff of the trial center through other alternative means (such as phone or virtual video). Details of adverse events and concomitant medications should be collected during communication. During this period, participants may not be able to participate in the laboratory tests and clinical evaluations specified during the study visit, but all relevant information should be recorded in detail. If laboratory data of subjects is collected or clinical evaluations are conducted through alternative methods, relevant information should be recorded in detail.

Primary outcome measures: Safety indicators

1. Demography/Medical History:

   i. Present medical history: including diagnostic basis, related symptoms, developmental history, current and past medication/recovery treatment status, etc; ii. History of other internal or surgical diseases (especially drug allergies, spinal trauma, etc.); iii. Abnormalities in gestational age and prenatal examinations; iv. Previous hospitalizations since birth, including duration of hospitalization, reasons, treatment received, and disease progression; If feasible, provide ICD-10 coding information for each hospitalization diagnosis; v. Family history
2. Physical examination:

   i. Genernal physical examination including neurological examination must be performed and recorded at designated visits, which should include at least the following contents: head/neck, eyes, ears, nose/throat, cardiovascular system, lungs, abdomen, musculoskeletal system, central nervous system, and skin.

   ii. Vital signs, height, and weight: Before measuring vital signs, subjects should rest in a quiet and undisturbed environment for at least 3 minutes, including body temperature, systolic and diastolic blood pressure, respiratory rate, pulse, and blood oxygen saturation.

   iii. After intrathecal injection of AAV-MECP2, lie flat for 6 hours with the pillow removed, and measure and record blood pressure, respiratory rate, pulse, and oxygen saturation every 15 minutes (± 5 minutes)in the first 2 hours; Afterwards, monitor the above indicators every hour (± 15 minutes) until 6 hours after intrathecal injection of AAV-MECP2.

   iv. During the screening period, height needs to be measured and weight measured at designated visits.
3. Laboratory investigations： i. Urine routine: color, specific gravity, pH value, glucose, protein, blood, ketone bodies, bilirubin, urobilinogen, nitrite, leukocyte esterase (test paper method), microscopic examination (if blood or protein test results are abnormal).

   ii. Blood routine: red blood cell count, hemoglobin, platelet count, white blood cell count and classification count, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin concentration, and reticulocyte count; iii. Morphological Examination of red Cells iv. Blood biochemistry: aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transferase (GGT), alkaline phosphatase (ALP), total bilirubin, direct bilirubin, total protein, creatinine, urea nitrogen, potassium, sodium, and calcium.

   v. Blood glucose and glycosylated hemoglobin; vi. The myocardial enzyme spectrum: creatine kinase (CK), creatine kinase isoenzyme (CK-MB), hydroxybutyrate dehydrogenase (HBDH), lactate dehydrogenase (LDH), and high-sensitivity troponin I (hsTnI).

   vii. The coagulation function: activated partial thromboplastin time (APTT), prothrombin time (PT), thrombin time (TT), fibrinogen (Fg, FIB), and D-dimer.

   viii. Immune function: peripheral blood lymphocyte subpopulation count:% CD3、%CD4、% CD8、CD4/CD8、%CD19、%CD16CD56； Complement system: Total complement activity (CH50), C3 activity and quantification, C4 activity and quantification.

   ix. Serum cytokines include: TNFα、IFN-γ、IL-10. x. Plasma ADAMTS13 factor and inhibitor. xi. Serum AAV9 neutralizing antibody.
4. Electrocardiogram (ECG): A conventional 12 lead ECG is obtained using an ECG device that can automatically calculate heart rate and measure PR, QRS, QT, and QTc intervals.
5. Echocardiography: During the screening period, a transthoracic color echocardiography examination will be scheduled to rule out potential cardiac lesions and cardiac dysfunction. The examination was interpreted and analyzed by ultrasound doctors and cardiologists at the research center.
6. Chest X-ray: During the screening period, chest X-ray examination is mainly conducted to exclude pulmonary infections that frequently occur in patients. If it is difficult to make a clear diagnosis on plain film, with the consent of the subject's guardian, an additional chest CT plain scan can be performed.
7. Head MRI: During the screening period, a head MRI plain scan is required to detect any anatomical abnormalities or other central nervous system lesions that need to be excluded. Two head MRI scans scheduled during the follow-up period were used to evaluate the toxicity associated with AAV-MECP2 injection and monitor central nervous system development.

Secondary outcome measures: Efficacy evaluation

1. RTT Specific Clinical Global Impressions Scale Severity (CGI-S) and Clinical Global Impressions Scale Improvement (CGI-I);
2. Rett Severity Assessment Questionnaire (RSSS);
3. Rett Syndrome Behavior Questionnaire (RSBQ);
4. Revised Motor Behavior Assessment (R-MBA);
5. Rett Syndrome Hand Function Scale (RSHFS);
6. Children's Sleep Habits Questionnaire;
7. Rett Parenting Stress Questionnaire;
8. Griffiths Developmental Rating Scale - Chinese Version (GDS-C): Only relative developmental age is used as the validity evaluation. If the age is over 8 years old and the ability is under 6 years old, GDS-C evaluation is still used;
9. Autism Diagnosis Behavior Observation Scale (ADOS);
10. Adaptive Behavior Assessment Scale for Children Aged 0-6 (Second Edition) - Parent Assessment Form;
11. Aberrant Behavior Scale (ABC);
12. Repetitive Stereotyped Behavior Scale-Revised (RBS-R);
13. Video evidence: Short video recordings will be made of the evaluation process of the subjects during the baseline period, medication hospitalization period, and 1, 3, 6, and 12 months after injection. If abnormal behavior occurs at other times, researchers may also decide to add video evidence. Parents/legal guardians can also provide home videos with improved display functions. After the recording is completed, the research team will immediately upload the video to an encrypted computer or laptop and delete the video file from the camera storage card. Any video received by the cooperating party will be considered confidential research data. The research team and partners will be responsible for protecting the identity information of the subjects and their parents/guardians in the video recording;
14. Electroencephalogram (EEG);
15. Wearable wristband: record sleep conditions;
16. Epilepsy records: During the study, subject guardians were required to record the occurrence of seizures, including all dates with and without seizures, including the presentation, duration, frequency, and date of seizures. Carry it with you at each follow-up visit for researchers to assess the frequency and duration of epileptic seizures.

The frequency of epileptic seizures will be defined using ordered variables with five categories: increase, no change, 75% remission, 50% remission, and no seizures.

Immunogenicity assessment:

In order to alleviate the immune response of the body to AAV gene therapy drugs, subjects need to take prophylactic oral corticosteroids and use prednisolone 24 hours before receiving injection. The dosage of prednisolone decreased gradually, and the medication time was not less than 2 months.

During the use of glucocorticoids, regular liver function check ups should be conducted to determine whether medication can be reduced or stopped based on liver function indicators. If the GGT, AST, or ALT values are ≥ 2 × ULN, researchers need to provide corresponding treatment based on the individual situation of the subjects. Based on previous clinical experience with AAV drug use, the high-risk period for liver enzyme rebound is within 2 weeks of hormone reduction or discontinuation. Therefore, liver function monitoring should be strengthened during this stage. For the above-mentioned prednisolone use and reduction plan, researchers can make personalized adjustments based on the safety assessment of the subjects. In addition to liver function, monitoring results of peripheral blood antigen-specific T cells may also need to be considered, and other immunosuppressive agents may be added if necessary. If the glucocorticoids used are preparations other than prednisolone, the dosage and withdrawal plan should be formulated based on the equivalent dose of prednisolone after conversion.

Informed consent:

Children under the age of 8 years participating in clinical trials should obtain a signed informed consent form from their guardian, and should be informed of relevant information about the clinical trial within the scope that the subjects can understand. When the child has the ability to make a decision to agree to participate in the clinical trial, their own consent should also be obtained; Children over 8 years old (including 8 years old) participating in clinical trials, if they have the ability to sign the informed consent form, both themselves and their guardians should sign the informed consent form. If they do not have the ability to sign the informed consent form, their guardians should sign the informed consent form.

Adverse medical events and treatments other than concomitant:

Medication/drugs that occur from the signing of the informed consent form until the first administration shall be recorded as medical history/comorbidities and treatment history in eCRF, and shall not be recorded on the AE page and concomitant medication/treatment page; Unless the injury/damage is caused by clinical laboratory examination procedures, it shall be recorded as an AE on the AE page, and for other treatments other than concomitant medication/drugs for this AE, they shall be recorded on the concomitant medication/treatment page accordingly.

The specific technical route is detailed in the research schedule.

Expected adverse reactions and treatment methods:

The risks associated with participants in this study mainly include risks related to drug administration procedures (sheath puncture), risks related to the investigational drug AAV-MECP2, and risks related to prophylactic immunosuppression.

Risks associated with sheath injection puncture:

1) Sheath injection puncture is generally considered safe, and the selected subjects will undergo a head magnetic resonance imaging (MRI) scan before lumbar puncture to rule out the possibility of intracranial space occupying lesions (especially in the posterior fossa) or increased intracranial pressure. The possible risks of lumbar puncture include the following: i. Headache after lumbar puncture: Patients undergoing lumbar puncture experience headaches due to fluid infiltration into nearby tissues after puncture. Headaches usually start within a few hours to two days after surgery and may be accompanied by nausea, vomiting, and dizziness. Headaches usually occur while sitting or standing, and can be relieved when lying down. Headaches after lumbar puncture may last for several hours to a week or longer.

ii. Discomfort or pain in the back: There may be pain or tenderness in the lower back. The pain may spread to the back of the leg.

iii. Bleeding: Bleeding near the puncture site, or in rare cases, it may occur in the epidural space.

The administration of drugs in this study was carried out by qualified doctors in the hospital treatment room. Before injection, the injection area was disinfected and covered with cloth. After injection, disinfection and compression hemostasis were performed, and the patient was bedridden for 6 hours with the pillow removed. After surgery, the subjects will be closely monitored to ensure that any possible complications are detected and treated in a timely manner.

Risks associated with AAV-MECP2:

The subject may experience allergic reactions to AAV-MECP2. Due to the immune response induced by intrathecal injection of AAV, subjects are usually unable to receive other gene therapies delivered by AAV vectors of the same serotype.

At present, there are three clinical trials (NCT05317780, NCT05419492, and NCT04833970) registered on the clinicaltrials.gov website for administering AAV drugs to the lateral ventricle for central nervous system diseases, but safety or efficacy clinical data have not yet been disclosed. AVXS-101 is the intrathecal version of the SMA gene therapy Zolgensma. A phase 1 dose escalation study conducted in subjects aged 6-60 months showed that AVXS-101 was safe and well tolerated when administered intrathecally at a maximum dose of 2.4 × 10^14 vg/person, with only one subject experiencing elevated transaminase levels without elevated bilirubin; One subject experienced thrombocytopenia (count below 75 × 10^9/L), which resolved spontaneously without intervention.

The following summarizes the serious adverse reactions (events) reported in AAV drugs that have been marketed or in clinical trials:

1. Hepatotoxicity. Reported on intravenous injection of AAV drugs for the treatment of SMA, Duchenne muscular dystrophy (DMD), and X-linked myopathy (XLMTM). The occurrence of hepatotoxicity is significantly correlated with the dosage of the drug administered, and severe cases of hepatotoxicity are only seen in subjects receiving AAV doses > 5 × 10^13 vg. Except for the liver toxicity in XLMTM, which is considered to be related to the patient's underlying liver disease, the published mechanism of other liver toxicity cases is considered to be liver cell injury mediated by CD8+T cells targeting AAV.
2. Thrombotic microvascular disease. Reported in the treatment of SMA and DMD with intravenous injection of AAV drugs, the occurrence of this event is also dose-dependent, and all cases were subjects who received AAV doses ≥ 5 × 10^13 vg. Due to the presence of laboratory evidence of complement activation in many of these cases, it is considered that their occurrence is related to the activation of the complement system by antigen antibody complexes targeting AAV. The cases generally occur within 1-2 weeks after infusion, and are characterized by thrombocytopenia, microangiopathic hemolytic anemia and acute kidney injury. Symptoms include vomiting, hypertension, oliguria/anuria, edema. If the following conditions occur after medication, thrombotic microangiopathy should be considered: platelet count below 50 ×10^9/L or a progressive decrease of ≥ 50%; accompanied by hemolytic anemia (hemoglobin reduction of ≥ 2 g compared to before medication, increase in lactate dehydrogenase and total bilirubin and indirect bilirubin compared to before medication); increased reticulocytes; acute kidney injury; in addition, other laboratory tests show elevated serum creatinine, proteinuria or hematuria. Once these conditions are found, timely treatment is required.
3. Myocarditis and myositis. Only reported on intravenous injection of AAV drugs in DMD. Based on the specific DMD gene mutation pattern, onset time, and response to immunosuppressive therapy present in the case, it is speculated that the essence of such toxic events is the immune response of the body to the genetically modified product "mini anti muscle atrophy protein".
4. Dorsal root ganglion (DRG) toxicity. The toxicity of DRG with clinical manifestations (abnormal hand and foot sensation) has only been reported in one patient with familial lateral sclerosis (ALS). This case received an intrathecal dose of 4.2 × 10^14 vg of AAV drug. The toxicity of DRG reported in other studies was accidentally discovered during the autopsy of AAV drug subjects, and the subjects had no relevant clinical manifestations before their death.
5. Abnormal brain MR signals. A clinical trial was reported on the treatment of late infantile Batten disease (CLN2 disease) by bilateral brain parenchymal injection of AAV drugs under stereotaxic localization. Within 48 hours after injection, the subject's head brain MR showed T2 hyperintensities, diffusion-weighted hyperintensities, and diffusion limited signals localized to the injection site. Subsequent MR follow-up showed that all subjects developed new T2 high signal areas. The researchers did not find any clinical sequelae associated with abnormal MR signals. It is speculated that the abnormal MR signals that appear early after administration are related to the sustained tissue edema/inflammation caused by the highest concentration of AAV drugs around the injection catheter tip, while the T2 high signals that appear later are difficult to determine whether they are related to disease progression, AAV drugs, or injection procedures.

Studies on patient samples (1 year after administration) and non-human primates (1 month after injection) have shown that the likelihood of AAV integration into the genome is low. Based on the safety record of AAV in clinical trials, the current consensus in the field of gene therapy is that AAV has low genetic toxicity in humans.

Preliminary preclinical safety evaluations of AAV-MECP2 in humanized RTT mice and crab eating macaques showed that, AAV-MECP2 did not cause liver or kidney function damage, nerve damage, immune toxicity, or histopathological changes in important organs in animals, and the general condition of the animals was good. Therefore, the existing data of AAV-MECP2 does not indicate clear clinical risks. The most common adverse event expected for subjects receiving AAV-MECP2 may be grade 1/2 elevation of liver enzymes.

Risks associated with preventive immunosuppression:

This protocol stipulates that starting from one day before AAV-MECP2 administration, oral administration of 1 mg/kg prednisolone or equivalent dose of other glucocorticoids should be started. The dosage of prednisolone decreased gradually, and the medication time was not less than 2 months. The purpose of using glucocorticoids is to suppress the innate and acquired immune responses induced by AAV vectors, and reduce immune reactions that are detrimental to safety and efficacy. When using hormones, adverse events related to hormones, including opportunistic infections, will be monitored in the subjects.

Corticosteroids (such as methylprednisolone and prednisone) have several clear side effects, including hypertension, tachycardia, congestive heart failure, changes in serum electrolytes, hyperglycemia, pain, elevated urea nitrogen and creatinine, osteoporosis and ischemic necrosis, decreased anti infective ability, dizziness, tremors, emotional instability, insomnia, nausea, vomiting, weight gain, elevated intraocular pressure, and the induction of cataracts.

During the use of hormones, researchers will closely monitor the above-mentioned adverse events, especially opportunistic infections that may occur in the subjects.

Statistical analysis:

This study is an early dose exploration study with the main objective of evaluating safety, therefore no formal sample size calculation was conducted.

The safety and tolerability of treatment are evaluated based on the frequency and severity of adverse events occurring within one year after administration. The proportion of subjects with any AE, any SAE, any AE related to the investigational drug, and any ≥ grade 3 AE will be statistically analyzed as a whole and by System Organ Classes (SOC) and preferred term (PT), respectively. The incidence of adverse events in different dose cohorts will also be statistically analyzed separately.

Due to the small sample size and the possibility of varying effectiveness indicators among subjects at different disease stages, all efficacy analyses in this study are descriptive and do not involve inferential statistics.

ELIGIBILITY:
Inclusion Criteria:

1. 4-10 years old (at the time of signing the informed consent form), female, who meets the typical RTT diagnosis criteria in 2010.
2. Gene testing confirms functional loss mutations in the MECP2 gene.
3. Complete all Class I vaccination required by the national regulations before the age of enrollment, and the final dose of vaccination must be completed at least 42 days before enrollment.
4. Participate in this study with the informed consent of the guardian, understand the risks of intrathecal injection procedures, and agree to collect blood, urine, and cerebrospinal fluid biological samples required for the experiment, as well as receive necessary blood or blood product treatment or other necessary medical treatment if necessary for the condition.

Exclusion Criteria:

1. Suffering from neurodevelopmental disorders other than MECP2 gene functional loss mutations, or pathogenic gene mutations other than MECP2 gene functional loss mutations discovered by whole exome sequencing.
2. Abnormal neurological function caused by traumatic brain injury or suffocation and hypoxia.
3. Through MRI scan, brain tumors or intracranial space-occupying lesions are detected.
4. Comprehensive abnormal psychomotor development has occurred within 6 months after birth.
5. Diagnosed as atypical RTT.
6. Has MECP2 gene mutation, but clinical diagnosis does not match RTT.
7. Need invasive respiratory support.
8. There are contraindications for lumbar puncture or intrathecal injection, including high cerebrospinal fluid pressure, obvious skin infection at the puncture site, trauma, epidural abscess, severe spinal lesions, deformities, spinal cord compression, bleeding tendency (bleeding tendency caused by the use of heparin, warfarin, etc.
9. Have experienced status epilepticus (> 30 minutes) or recurrent unstable seizure control (> 2 generalized seizures per week) in the past 3 months.
10. In addition to RTT, there are other unstable systemic diseases, including active bacteria, fungi, or HIV, hepatitis A, hepatitis B infection.
11. There are significant laboratory indicators with abnormalities: any detection value of alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyltransferase (GGT), alkaline phosphatase (ALP) is ≥ 2 times the upper limit of normal (ULN).
12. Total bilirubin ≥ 1.5 × ULN.
13. Creatinine ≥ 159 μ mol/L.
14. Hemoglobin (Hb) < 80 g/L.
15. Prothrombin time (PT) prolonged by ≥ 3 seconds.
16. Prolonged activated partial thromboplastin time (APTT) by ≥ 10 seconds.
17. Fasting blood glucose ≥ 7.0 mmol/L.
18. HbA1c ≥ 6.5%.
19. Platelet values are outside the range of 100-300 ×10^9/L.
20. Serum anti AAV neutralizing antibody titer > 1:50 (ELISA immunoassay).
21. Systemic use of immunosuppressive drugs (cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immune globulin, and rituximab) other than protocol-specified prophylaxis within 3 months prior to enrollment.
22. Previously received gene therapy.
23. Plan to make changes in clinical medication during this clinical trial, participate in other clinical trials, or have received other investigational drug treatments within 30 days or 5 half lives (whichever is longer) before enrollment.
24. Known allergy to investigational drug.
25. Any condition that, in the opinion of the Investigator, patients are not appropriate to participate in the study.

Ages: 4 Years to 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2029-10-23 (Estimated); Study Completion 2029-10-23 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | Baseline through week 52
  Incidence of drug-related adverse events (AEs) and serious adverse events (SAEs), assessed through medical history, physical exams, vital signs, laboratory tests (blood/urine), ECG, echocardiography, chest X-ray, and head MRI.

SECONDARY OUTCOMES:
Exploratory Efficacy | Baseline through week 52
  Change from baseline in disease severity as assessed by the Rett Syndrome Clinical Global Impressions-Severity (CGI-S). This 7-point clinician-administered scale (1 = normal, 7 = extremely ill) evaluates overall disease severity; higher scores indicate greater severity.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in clinical improvement as assessed by the Rett Syndrome Clinical Global Impressions-Improvement (CGI-I). This 7-point clinician-administered scale (1 = very much improved, 7 = very much worse) measures global functional changes; higher scores indicate worsening.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in disease severity as assessed by the Rett Severity Assessment Scale (RSSS). This clinician-rated scale evaluates clinical features across multiple domains (motor, respiratory, behavioral); higher scores correlate with greater severity.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in behavioral symptoms as assessed by the Rett Syndrome Behavior Questionnaire (RSBQ). This 45-item caregiver-reported questionnaire (scores 0-2 per item) measures mood, breathing abnormalities, anxiety, and motor function; higher scores indicate greater severity.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in motor function as assessed by the Revised Motor Behavior Assessment (R-MBA). This clinician-administered 34-item scale (scores 0-4 per item) evaluates daily activities (behavioral/social, respiratory, motor); higher scores reflect greater impairment.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in hand function as assessed by the Rett Syndrome Hand Function Scale (RSHFS). This clinician-rated tool measures fine motor skills and hand stereotypies; higher scores indicate poorer function.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in sleep quality as assessed by the Children's Sleep Habits Questionnaire. This caregiver-reported tool evaluates sleep duration, disturbances, and patterns; higher scores indicate worse sleep.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in developmental level as assessed by the Griffiths Developmental Scale-Chinese Version (GDS-C). This clinician-administered scale measures developmental milestones across domains (locomotion, social-emotional, etc.); higher scores indicate better function.Change from baseline in developmental level as assessed by the Griffiths Developmental Scale-Chinese Version (GDS-C). This clinician-administered scale measures developmental milestones across domains (locomotion, social-emotional, etc.); higher scores indicate better function.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in autism-related behaviors as assessed by the Autism Diagnostic Observation Scale (ADOS). This clinician-administered tool evaluates social communication and repetitive behaviors; higher scores indicate greater impairment.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in behaviors as assessed by the Abberant Behavior Checklist (ABC). This Parent-administered Checklist evaluates behaviors across the domains (irritability, lethargy, stereotypy etc.); higher scores indicate greater impairment.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in behaviors as assessed by Repetitive Stereotyped Behavior Scale-Revised (RBS-R). This 3-point Parent-administered scale (0 = normal, 3 = extremely impairment) evaluates repetitive stereotyped behaviors; higher scores indicate greater impairment.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in Adaptive ability by Behavior Assessment Scale for Children Aged 0-6 (Second Edition) (ABAS-II) - Parental Assessment Form. This Parent-administered Checklist evaluates behaviors across the domains (social communication, locomotion, self-care skill etc.); higher scores indicate better function.
Exploratory Efficacy | Baseline through week 52
  Change from baseline in Parenting Stress by Parenting Stress Questionnaire (PSQ). PSQ typically consists of 34 items rated on a 4-point Likert scale (1 = Strongly Disagree to 4 = Strongly Agree). Total scores range from 34 to 136, calculated by summing all item responses. Higher scores indicate greater parenting stress.
Exploratory Efficacy | Baseline through week 52
  Epilepsy Record: during the study, epileptic subject guardians were required to record seizures, including all dates with and without seizures, including the presentation, duration, frequency, and date of seizures; The frequency of epileptic seizures will be defined using ordered variables with five categories: increase, no change, 75% remission, 50% remission, and no seizures.
Exploratory Efficacy | Baseline through week 52
  Video evidence: Short video recordings will be made of the evaluation process of the subjects during the baseline period, medication hospitalization period, and 1, 3, 6, and 12 months after injection. If abnormal behavior occurs at other times, researchers may also decide to add video evidence
Exploratory Efficacy | Baseline through week 52
  Change from baseline in Changes in neurophysiology by video electroencephalogram
Exploratory Efficacy | Baseline through week 52
  Change from baseline in sleep status via wearable wristband to record sleep conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Ask the organization ethic committee for Primary data when publishing or after published paper.